CLINICAL TRIAL: NCT03922022
Title: Exercise is Medicine for Chronic Diseases: a Pilot Study for Future Randomized Controlled Trial
Brief Title: Exercise is Medicine: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTEC-2019-0121
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Intervention Model Description: patients will go to different classes: (i) Hypertension basic exercise class (ii) Hypertension advanced exercise class (iii) diabetes basic exercise class (iv) diabetes advanced exercise class; if the patient has normal BMI AND reported some regular exercise, they will be prescribed the advanced level class. There is no control group for this pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIM group (Experimental): patients will go to different classes: (i) Hypertension basic exercise class (ii) Hypertension advanced exercise class (iii) diabetes basic exercise class (iv) diabetes advanced exercise class; if the patient has normal BMI AND reported some regular exercise, they will be prescribed the advanced level class. There is no control group for this pilot study
  Interventions: Behavioral: EIM exercise classes and intervention

INTERVENTIONS:
Behavioral: EIM exercise classes and intervention — This is a complex intervention. On recruitment, they will be seen by a nurse and counselled using motivational technique. They will then undergo a 12-week class. The exercise levels will be regularly feedback to the patients by use of mobile devices and trackers. Peer support is formed during the 12-week class. Resources to continue exercise will be provided to patients. Regular monitoring of physical improvement will be feedback to patients to encourage continued exercise.

SUMMARY:
Background: Regular exercise is beneficial to patients with hypertension and/or diabetes mellitus. However, most patients cannot maintain exercise habit. The investigators had developed a program called the "exercise is medicine"(EIM), combining motivational technique, information technology use and teaching exercise techniques. Before using this intervention in a main randomized controlled trial, the investigators would like to test its feasibility and acceptability. It is hypothesized that this program is feasible and acceptable to patients.

Method: 40 patients with HT and/or DM will be recruited to attend the EIM intervention. Primary outcomes will be the rate of recruitment and rate of retention. Other clinical outcomes will be obtained before and immediately after the 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* clinic systolic BP(SBP) higher than 130mmHg (for HT class) because the Hong Kong primary care office guideline, as of Jan 2019, regarded good control of SBP to be ≤130mmHg, OR HbA1c >7% (for DM class)
* self-reported regular exercise of ≤3 times per week - this cut-off is arbitrary but people who exercise more than 3 times may have little space for improvement; and these patients will unlikely be referred to EIM when it is implemented in routine clinical practice, - who have used any mobile apps on their phone (because the intervention involve use of apps to monitor and remind regular exercise)

Exclusion Criteria:

* patients with diagnosed chronic obstructive lung disease and recent stroke (within last 12 months) are excluded because there are other evidence-proven and well-structured programmes for these patients in the Hospital Authority (HA), for instance, pulmonary rehabilitation program conducted by physiotherapy and/or occupational therapist in HA. - - acute myocardial infarction in last 6 months
* ongoing angina
* uncontrolled cardiac arrhythmia
* acute diseases including known active endocarditis/acute pulmonary embolism, pulmonary infarction, deep vein thrombosis, acute aortic dissection, acute myocarditis
* known aortic stenosis
* known heart failure
* known obstructive left main coronary artery stenosis
* uncontrolled ventricular rates
* complete heart block
* known hypertrophic obstructive cardiomyopathy
* mental impairment that limit co-operation
* resting blood pressure with systolic blood pressure >180mmHg or diastolic blood pressure >110mmHg
* known anaemia with haemoglobin level less than 11gm/dL
* known uncorrected electrolyte imbalance
* known uncontrolled hyperthyroidism.
* For DM patients, patients with proliferative diabetic retinopathy and recent retinal bleeding (in last 12 months) are also excluded due to reports that vigorous exercise may increase blood pressure and led to retinal bleeding in these patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
rate of retention | from recruitment to finish of the 12-week program
  rate of retention
Rate of recruitment | from recruitment to the start of the 12-week program
  Rate of recruitment

SECONDARY OUTCOMES:
Clinic blood pressure (BP) | on recruitment and after the 12- week class
  Clinical BP will be measured 3 times and the last 2 will be averaged
HbA1c (glycosylated hemoglobin) | on recruitment and after the 12- week class
  for DM patients only
Godin-Shephard Laiesure-Time Physical Activity Questoinnaire | on recruitment and after the 12- week class
  a validated questionnaire to detect change in exercise level
body mass index (BMI) | on recruitment and after the 12- week class
  the weight and height of the patients will be measured
body fat percentage | on recruitment and after the 12- week class
  body fat percentage
lipid level | on recruitment and after the 12- week class
  this will include low-density lipoprotein, high-density lipoprotein, and total lipoprotein
9-item patient health questionnaire | on recruitment and after the 12- week class
  a validated questionnaire to detect depressive symptoms
Generalized anxiety disorder-7 | on recruitment and after the 12- week class
  a validated questionnaire to detect anxiety symptoms
EQ-5D-5L | on recruitment and after the 12- week class
  a validated questionnaire to measure quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will make available on personal requests to investigators